CLINICAL TRIAL: NCT01570712
Title: Evaluation of the "Housing First Program" in Homeless Patients With Severe Mental Disorders in France: a Multicentric Randomized Controlled Study
Brief Title: Evaluation of the "Housing First Program" in Homeless Patients With Severe Mental Disorders in France
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2011-A00668-33; 2011-12 (Other: AP HM)
Record Dates: First submitted 2012-04-02; First posted 2012-04-04 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Subnormal; Mental, Severe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Housing First Program (Experimental)
  Interventions: Other: HOUSING FIRST PROGRAM
- traditional French services (Active Comparator)
  Interventions: Other: traditional French services

INTERVENTIONS:
Other: HOUSING FIRST PROGRAM — Realization of a psychosocial organic evaluation and a citizen;
  * Support in the development and the maintenance of the housing;
  * Support in the diverse steps (administrative, judicial, financiers, etc.);
  * Support around addictions / alcohol;
  * Supportin the family and social relations, in the environment of the person -to favor the occupational integration, by prioritizing the insertion in ordinary environment(middle)
  * to favor the access and the preservation of the patient to the psychiatric and somatic care, to the devices and the departments favoring the social insertion and the integration.
  Arms: Housing First Program
Other: traditional French services — The person will not receive from intervention of the team of site, but the person can resort(turn) without limitation to all the range of services said " about "common law " set up in the direction of the persons homeless persons, as well as to every type of care. She can too reach the housing and\or the restoring, but this by means of the existing devices
  Arms: traditional French services

SUMMARY:
As mental health care shifted from state psychiatric hospitals to the community in France and western countries, the mental health system became inevitably involved in housing as it strove to meet the broader psychosocial needs of consumers. Simultaneously, as many consumers found themselves unable to find stable living in the community and struggling with addictions, they became a significant subgroup within a larger homeless population, which has received increasing policy attention over the past three decades. There are two distinct service models for adults who have severe mental illness and are homeless: the residential continuum model and the Housing First model.

ELIGIBILITY:
Inclusion Criteria:

aged over 18;

* who are absolutely homeless or precariously housed. Absolutely homeless is defined as having had no fixed place to stay for at least the past seven nights with little likelihood of finding a place in the coming month. Precariously housed is defined as being housed a in single room occupancy, rooming house, or hotel/motel as a primary residence AND in the past year having experienced two or more episodes of being absolutely homeless OR one episode of being absolutely homeless that lasted for more than four weeks in the preceding 12 months.
* living with schizophrenia or bipolar disorder (diagnosis of DSM-IV);
* with a sufficient understanding of written and spoken French to be able to provide informed consent and to participate to face-to-face interviews;
* affiliated to a social protection;
* who have lived in the city targeted for at least 6 months and willing to stand in the city during the 2 next years;
* with a global score measured on Multnomah Community Ability Scale (MCAS) (scale <=62 (high need criteria));
* hospitalized at least twice on the past 12 months OR held in prison on the past 24 months OR presenting substance or alcohol abuse or dependence (high need criteria).

Exclusion Criteria:

* being considered unable to provide informed consent;
* having dependent children;
* pregnancy;
* or a DSM-IV Axis I diagnosis other than schizophrenia or bipolar disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2011-08; Primary Completion 2016-05 (Actual); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
healthcare utilisation | 3 YEARS
  hospitalizations, hospital days, and emergency department visits

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — Assistance Publique hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Loubiere S, Lemoine C, Boucekine M, Boyer L, Girard V, Tinland A, Auquier P; French Housing First Study Group. Housing First for homeless people with severe mental illness: extended 4-year follow-up and analysis of recovery and housing stability from the randomized Un Chez Soi d'Abord trial. Epidemiol Psychiatr Sci. 2022 Feb 7;31:e14. doi: 10.1017/S2045796022000026. PMID 35125129
- [Derived] Tinland A, Loubiere S, Cantiello M, Boucekine M, Girard V, Taylor O, Auquier P. Mortality in homeless people enrolled in the French housing first randomized controlled trial: a secondary outcome analysis of predictors and causes of death. BMC Public Health. 2021 Jul 2;21(1):1294. doi: 10.1186/s12889-021-11310-w. PMID 34215235
- [Derived] Loubiere S, Tinland A, Taylor O, Loundou A, Girard V, Boyer L, Auquier P. Determinants of healthcare use by homeless people with schizophrenia or bipolar disorder: results from the French Housing First Study. Public Health. 2020 Aug;185:224-231. doi: 10.1016/j.puhe.2020.05.019. Epub 2020 Jul 14. PMID 32679400
- [Derived] Fond G, Boyer L, Boucekine M, Girard V, Loubiere S, Lenoir C, Auquier P, Tinland A; French Housing First Study Group. Illness and drug modifiable factors associated with violent behavior in homeless people with severe mental illness: results from the French Housing First (FHF) program. Prog Neuropsychopharmacol Biol Psychiatry. 2019 Mar 2;90:92-96. doi: 10.1016/j.pnpbp.2018.11.006. Epub 2018 Nov 10. PMID 30423419
- [Derived] Rhenter P, Tinland A, Grard J, Laval C, Mantovani J, Moreau D, Vidaud B, Greacen T, Auquier P, Girard V. Problems maintaining collaborative approaches with excluded populations in a randomised control trial: lessons learned implementing Housing First in France. Health Res Policy Syst. 2018 Apr 19;16(1):34. doi: 10.1186/s12961-018-0305-1. PMID 29673362
- [Derived] Tinland A, Zemmour K, Auquier P, Boucekine M, Girard V, Loubiere S, Fond G, Boyer L; French Housing First Study Group. Homeless women with schizophrenia reported lower adherence to their medication than men: results from the French Housing First experience. Soc Psychiatry Psychiatr Epidemiol. 2017 Sep;52(9):1113-1122. doi: 10.1007/s00127-017-1411-z. Epub 2017 Jun 27. PMID 28656452
- [Derived] Tinland A, Fortanier C, Girard V, Laval C, Videau B, Rhenter P, Greacen T, Falissard B, Apostolidis T, Lancon C, Boyer L, Auquier P. Evaluation of the Housing First program in patients with severe mental disorders in France: study protocol for a randomized controlled trial. Trials. 2013 Sep 24;14:309. doi: 10.1186/1745-6215-14-309. PMID 24063556